CLINICAL TRIAL: NCT04380701
Title: A Multi-site, Phase I/II, 2-Part, Dose-Escalation Trial Investigating the Safety and Immunogenicity of Four Prophylactic SARS-CoV-2 RNA Vaccines Against COVID-19 Using Different Dosing Regimens in Healthy and Immunocompromised Adults
Brief Title: A Trial Investigating the Safety and Effects of Four BNT162 Vaccines Against COVID-19 in Healthy and Immunocompromised Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT162-01; 2020-001038-36 (EudraCT Number); U1111-1249-4220 (Other: WHO UTN)
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-01

CONDITIONS: Infections, Respiratory; Virus Diseases; Infection Viral; Vaccine Adverse Reaction; RNA Virus Infections; Protection Against COVID-19 and Infections With SARS CoV 2
Keywords: SARS-CoV-2; Severe Acute Respiratory Syndrome (SARS); Coronavirus Disease 2019; COVID-2019; Virus Diseases
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases; RNA Virus Infections; Severe Acute Respiratory Syndrome; COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- BNT162a1 (P/B) - Part A 18-55 years of age (Experimental): Escalating dose levels
  Interventions: Biological: BNT162a1
- BNT162b1 (P/B) - Part A 18-55 years of age (Experimental): Escalating dose levels
  Interventions: Biological: BNT162b1
- BNT162b2 (P/B) - Part A 18-55 years of age (Experimental): Escalating dose levels
  Interventions: Biological: BNT162b2
- BNT162c2 (P/B) - Part A 18-55 years of age (Experimental): Escalating dose levels
  Interventions: Biological: BNT162c2
- BNT162c2 (prime only) - Part A 18-55 years of age (Experimental): Single dose
  Interventions: Biological: BNT162c2
- BNT162b1 (P/B) - Part A 56-85 years of age (Experimental): Escalating dose levels
  Interventions: Biological: BNT162b1
- BNT162b2 (P/B) - Part A 56-85 years of age (Experimental): Escalating dose levels
  Interventions: Biological: BNT162b2
- BNT162b2 (P/B) - Part A 18-85 years of age (Expansion cohorts 11 to 13) (Experimental): Fixed doses used; cohort 11: alternative posology dose group expansion cohort; cohort 12: adaptive immune response dose group expansion cohort; cohort 13: immunocompromised (IC) participants expansion cohort
  Interventions: Biological: BNT162b2
- BNT162b2 (P/B) - Part A 18-85 years of age (Expansion cohort 14) (Experimental): fixed doses used; B-cell immune response dose group expansion cohort
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BNT162a1 — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: BNT162a1 (P/B) - Part A 18-55 years of age
Biological: BNT162b1 — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: BNT162b1 (P/B) - Part A 18-55 years of age; BNT162b1 (P/B) - Part A 56-85 years of age
Biological: BNT162b2 — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: BNT162b2 (P/B) - Part A 18-55 years of age; BNT162b2 (P/B) - Part A 18-85 years of age (Expansion cohort 14); BNT162b2 (P/B) - Part A 18-85 years of age (Expansion cohorts 11 to 13); BNT162b2 (P/B) - Part A 56-85 years of age
Biological: BNT162c2 — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: BNT162c2 (P/B) - Part A 18-55 years of age; BNT162c2 (prime only) - Part A 18-55 years of age

SUMMARY:
Originally, the study was planned to include two parts, i.e., Part A and Part B, however Part B was cancelled due to changes in the overall clinical development plan. The objectives originally described for Part B have been implemented in the ongoing development via a pivotal Phase I/II/III trial BNT162-02/C4591001 (ClinicalTrials.gov NCT: 04368728).

The conducted Part A was a dose-finding part to investigate the optimal dose of four different vaccines (BNT162a1, BNT162b1, BNT162b2, and BNT162c2), allowing dose adjustments upwards and downwards in younger participants. Doses tested in older participants and expansion cohorts were chosen based on acceptability of dosing in younger participants.

The vaccines BNT162a1, BNT162b1, BNT162b2, and BNT162c2 were administered using a Prime/Boost (P/B) regimen with two doses given ~21 days apart. The vaccine BNT162c2 was also administered using a Single dose (SD) regimen. Four additional expansion cohorts (cohorts 11, 12, 13, and 14) aged from 18 to 85 years received BNT162b2 using a P/B regimen only. In cohort 11, participants received BNT162b2 using one 3 μg prime dose (Dose 1) and one 30 μg boost dose (Dose 2) of BNT162b2. Participants in cohorts 12, 13, and 14 received two doses of BNT162b2 30 µg, each.

DETAILED DESCRIPTION:
This study was a multi-site, Phase I/II, open-label, dose-escalation study. The study included the first-in-human (FIH) dose and dose ranging groups for all four vaccines in healthy younger participants (aged 18 to 55 years [years]) and older participants (aged 56 to 85 years). The conducted Part A followed a dose escalation design. Discretionary dose de-escalation and refinement was also planned. Study participants with the FIH immunization and any subsequent dose escalation cohorts were immunized using a sentinel dosing/subject staggering. For any dose de-escalation or dose-refinement cohorts in younger adults, i.e., cohorts with doses lower than previously tested, participants were dosed using a subject staggering process. Cohorts in older participants were optional and dependent on acceptability of dosing in younger participants. Part A consisted of a treatment phase and a follow-up phase.

For the BNT162a1 3 µg arm, the Safety Review Committee (SRC) decided to stop dosing after 6 treated participants and to not administer the boost immunization (Dose 2). For the BNT162b1 60 µg arm, the SRC decided to not administer the boost immunization (Dose 2) for the 12 participants.

ELIGIBILITY:
Inclusion Criteria:

* Have given informed consent by signing the informed consent form (ICF) before initiation of any trial-specific procedures.
* They must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions (e.g., to practice social distancing and to follow good practices to reduce their chances of being infected or spreading COVID-19), and other requirements of the trial.
* They must be able to understand and follow trial-related instructions.
* For younger adult cohorts, volunteers must be aged 18 to 55 years, have a body mass index (BMI) over 19 kg/m^2 and under 30 kg/m^2, and weigh at least 50 kg at Visit 0. OR For older adult cohorts, volunteers must be aged 56 to 85 years, have a BMI over 19 kg/m^2 and under 30 kg/m^2, and weigh at least 50 kg at Visit 0. OR For the immunocompromised adult cohort (Cohort 13), volunteers must be aged 18 to 85 years, have a BMI over 19 kg/m^2 and under 30 kg/m^2, and weigh at least 50 kg at Visit 0.
* They must be healthy, in the clinical judgment of the investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs (systolic/diastolic blood pressure, pulse rate, body temperature, respiratory rate), and clinical laboratory tests (blood chemistry, hematology, and urine chemistry) at Visit 0. Note: Healthy volunteers with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included. OR For the immunocompromised cohort (Cohort 13); volunteers who have previously received solid organ transplant, or peripheral blood stem cell transplantation ≥6 months after transplantation, or individuals with human immunodeficiency virus (HIV) infection with a CD4+ T-cell count of ≥200 x 10^6 /L at Visit 0. Individuals with lower T-cell counts will be excluded from the trial on the basis that this represents a significant medical complication. In the clinical judgment of the investigator, volunteers must be immunocompromised but otherwise healthy. After consultation with the Medical Monitor, this may include individuals receiving immunosuppressant therapy due to another confounding disease at least 2 weeks prior to enrollment and/or at least 6 weeks following immunization with BNT162b2, and/or individuals with immunosuppressive treatment of an autoimmune disease if the disease is stable.
* Women of childbearing potential (WOCBP) must have a negative beta-human chorionic gonadotropin urine test at Visit 0 and Visit 1. Women that are postmenopausal or permanently sterilized will be considered as not having reproductive potential.
* WOCBP must agree to practice a highly effective form of contraception during the trial, starting after Visit 0 and continuously until 60 days after receiving the last immunization. WOCBP must agree to require their male partners to use condoms during sexual contact (unless male partners are sterilized or infertile).
* WOCBP must confirm that they practice at least one highly effective form of contraception for the 14 days prior to Visit 0.
* WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting after Visit 0 and continuously until 60 days after receiving the last immunization.
* Men who are sexually active with a WOCBP and have not had a vasectomy must agree to practice a highly effective form of contraception with their female partner of childbearing potential during the trial, starting after Visit 0 and continuously until 60 days after receiving the last immunization.
* Men must be willing to refrain from sperm donation, starting after Visit 0 and continuously until 60 days after receiving the last immunization.
* They must have confirmation of their health insurance coverage prior to Visit 0.
* They must agree to not be vaccinated during the trial, starting after Visit 0 and continuously until 28 days after receiving the last immunization.

Exclusion Criteria:

* Have had any acute illness, as determined by the investigator, with or without fever, within 72 hours prior to the first immunization. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the investigator, the residual symptoms will not compromise their well-being if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Are breastfeeding on the day of Visit 0 or who plan to breastfeed during the trial, starting after Visit 0 and continuously until at least 90 days after receiving the last immunization.
* Have a known allergy, hypersensitivity, or intolerance to the planned investigational medicinal product (IMP) including any excipients of the IMP.
* Had any medical condition or any major surgery (e.g., requiring general anesthesia) within the past 5 years which, in the opinion of the investigator, could compromise their well-being if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Have any surgery planned during the trial, starting after Visit 0 and continuously until at least 90 days after receiving the last immunization.
* Had any chronic use (more than 21 continuous days) of any systemic medications, including immunosuppressant's or other immune-modifying drugs (except for Cohort 13), within the 6 months prior to Visit 0 unless in the opinion of the investigator, the medication would not prevent, limit, or confound the protocol-specified assessments or could compromise subject safety. Note: Healthy volunteers with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.
* Had any vaccination within the 28 days prior to Visit 0.
* Had administration of any immunoglobulins and/or any blood products within the 3 months prior to Visit 0.
* Had administration of another investigational medicinal product including vaccines within 60 days or 5 half-lives (whichever is longer), prior to Visit 0.
* Have a known history of active or ongoing hepatitis B or hepatitis C infection; or except for Cohort 13: HIV-1 or HIV-2 infection within the 30 days prior to Visit 0.
* Have a positive polymerase chain reaction (PCR)-based test for SARS-CoV-2 within the 30 days prior to Visit 1.
* Have a positive drugs of abuse (for amphetamines, benzodiazepines, barbiturates, cocaine, cannabinoids, opiates, methadone, methamphetamines, phencyclidine, and tricyclic antidepressants) result at Visit 0 or Visit 1.
* Have a positive breath alcohol test at Visit 0 or Visit 1.
* Previously participated in an investigational trial involving lipid nanoparticles.
* Are subject to exclusion periods from other investigational trials or simultaneous participation in another clinical trial. When entering the follow-up phase, i.e., after completing the end of treatment (EoT) visit, subjects are allowed to participate in other clinical trials not investigating COVID-19 vaccines or treatments; subjects immunized with BNT162 vaccines in this clinical trial are allowed to participate in other clinical trials involving immunization with BNT162b2.
* Have any affiliation with the trial site (e.g., are close relative of the investigator or dependent person, such as an employee or student of the trial site).
* Have a history (within the past 5 years) of substance abuse or known medical, psychological, or social conditions which, in the opinion of the investigator, could compromise their well-being if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
* Have a history of hypersensitivity or serious reactions to previous vaccinations.
* Have a history of Guillain-Barré Syndrome within 6 weeks following a previous vaccination.
* Have a history of narcolepsy.
* Have history of alcohol abuse or drug addiction within 1 year before Visit 0.
* (Except for Cohort 13) Have a history of or suspected immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination at Visit 0.
* Have any abnormality or permanent body art (e.g., tattoo) that, in the opinion of the investigator, would obstruct the ability to observe local reactions at the injection site.
* Have had any blood loss >450 mL, e.g., due to donation of blood or blood products or injury, within the 7 days prior to Visit 0 or plan to donate blood during the trial, starting after Visit 0 and continuously until at least 7 days after receiving the last immunization.
* Have symptoms of COVID-19, e.g., respiratory symptoms, fever, cough, shortness of breath and breathing difficulties.
* Have had contact with persons diagnosed with COVID-19 or who tested positive for SARS-CoV-2 by any diagnostic test within the 30 days prior to Visit 1.
* Are soldiers, volunteers in detention, contract research organization (CRO) or sponsor staff or their family members.
* Regular receipt of inhaled/nebulized corticosteroids (except for Cohort 13).
* For older volunteers and for Cohort 13 only: Have a condition known to put them at high risk for severe COVID-19, including those with any of the following risk factors:
* Uncontrolled hypertension.
* Diabetes mellitus (HbA1c >8.5% ≥3 months, according to the medical history reported by the subject).
* Chronic obstructive pulmonary disease.
* Asthma.
* Chronic liver disease.
* Known Stage 3 or worse chronic kidney disease (glomerular filtration rate <60 mL/min/1.73 m^2); Except for post-renal transplant patients who should have (estimated) GFR ≥40 mL/min/1.73 m^2.
* Serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies.
* Sickle cell disease.
* Cancer (except for Cohort 13).
* Are immune compromised due to stem cell or organ-transplantation with significant medical complications such as acute or chronic graft rejection or graft versus host disease requiring intensive immunosuppressive treatment, transplant failure or infectious complications or other conditions that would be considered a contraindication for vaccination.
* Are immune compromised due to HIV infection with a CD4+ count of < 200 x 10^6 /L at screening or significant medical complications such as opportunistic infections, malignant complications (e.g., lymphoma, Kaposi sarcoma), other organ manifestations consistent with advanced AIDS or other conditions that would be considered a contraindication for vaccination.
* Resident in a long term facility.
* Current vaping or smoking (occasional smoking is acceptable).
* History of chronic smoking within the prior year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (5):
- Germany (5):
  - Contract Research Organization, Berlin
  - Universitäts Klinikum, Frankfurt am Main
  - Universitäts Klinikum, Heidelberg
  - Contract Research Organization, Kiel
  - Contract Research Organization, Mannheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muik A, Wallisch AK, Sanger B, Swanson KA, Muhl J, Chen W, Cai H, Maurus D, Sarkar R, Tureci O, Dormitzer PR, Sahin U. Neutralization of SARS-CoV-2 lineage B.1.1.7 pseudovirus by BNT162b2 vaccine-elicited human sera. Science. 2021 Mar 12;371(6534):1152-1153. doi: 10.1126/science.abg6105. Epub 2021 Jan 29. PMID 33514629
- [Background] Sahin U, Muik A, Derhovanessian E, Vogler I, Kranz LM, Vormehr M, Baum A, Pascal K, Quandt J, Maurus D, Brachtendorf S, Lorks V, Sikorski J, Hilker R, Becker D, Eller AK, Grutzner J, Boesler C, Rosenbaum C, Kuhnle MC, Luxemburger U, Kemmer-Bruck A, Langer D, Bexon M, Bolte S, Kariko K, Palanche T, Fischer B, Schultz A, Shi PY, Fontes-Garfias C, Perez JL, Swanson KA, Loschko J, Scully IL, Cutler M, Kalina W, Kyratsous CA, Cooper D, Dormitzer PR, Jansen KU, Tureci O. COVID-19 vaccine BNT162b1 elicits human antibody and TH1 T cell responses. Nature. 2020 Oct;586(7830):594-599. doi: 10.1038/s41586-020-2814-7. Epub 2020 Sep 30. PMID 32998157
- [Background] Sahin U, Muik A, Vogler I, Derhovanessian E, Kranz LM, Vormehr M, Quandt J, Bidmon N, Ulges A, Baum A, Pascal KE, Maurus D, Brachtendorf S, Lorks V, Sikorski J, Koch P, Hilker R, Becker D, Eller AK, Grutzner J, Tonigold M, Boesler C, Rosenbaum C, Heesen L, Kuhnle MC, Poran A, Dong JZ, Luxemburger U, Kemmer-Bruck A, Langer D, Bexon M, Bolte S, Palanche T, Schultz A, Baumann S, Mahiny AJ, Boros G, Reinholz J, Szabo GT, Kariko K, Shi PY, Fontes-Garfias C, Perez JL, Cutler M, Cooper D, Kyratsous CA, Dormitzer PR, Jansen KU, Tureci O. BNT162b2 vaccine induces neutralizing antibodies and poly-specific T cells in humans. Nature. 2021 Jul;595(7868):572-577. doi: 10.1038/s41586-021-03653-6. Epub 2021 May 27. PMID 34044428
- [Background] Vogel AB, Kanevsky I, Che Y, Swanson KA, Muik A, Vormehr M, Kranz LM, Walzer KC, Hein S, Guler A, Loschko J, Maddur MS, Ota-Setlik A, Tompkins K, Cole J, Lui BG, Ziegenhals T, Plaschke A, Eisel D, Dany SC, Fesser S, Erbar S, Bates F, Schneider D, Jesionek B, Sanger B, Wallisch AK, Feuchter Y, Junginger H, Krumm SA, Heinen AP, Adams-Quack P, Schlereth J, Schille S, Kroner C, de la Caridad Guimil Garcia R, Hiller T, Fischer L, Sellers RS, Choudhary S, Gonzalez O, Vascotto F, Gutman MR, Fontenot JA, Hall-Ursone S, Brasky K, Griffor MC, Han S, Su AAH, Lees JA, Nedoma NL, Mashalidis EH, Sahasrabudhe PV, Tan CY, Pavliakova D, Singh G, Fontes-Garfias C, Pride M, Scully IL, Ciolino T, Obregon J, Gazi M, Carrion R Jr, Alfson KJ, Kalina WV, Kaushal D, Shi PY, Klamp T, Rosenbaum C, Kuhn AN, Tureci O, Dormitzer PR, Jansen KU, Sahin U. BNT162b vaccines protect rhesus macaques from SARS-CoV-2. Nature. 2021 Apr;592(7853):283-289. doi: 10.1038/s41586-021-03275-y. Epub 2021 Feb 1. PMID 33524990
- [Background] Ji RR, Qu Y, Zhu H, Yang Y, Vogel AB, Sahin U, Qin C, Hui A. BNT162b2 Vaccine Encoding the SARS-CoV-2 P2 S Protects Transgenic hACE2 Mice against COVID-19. Vaccines (Basel). 2021 Apr 1;9(4):324. doi: 10.3390/vaccines9040324. PMID 33915773
- [Background] Li J, Hui A, Zhang X, Yang Y, Tang R, Ye H, Ji R, Lin M, Zhu Z, Tureci O, Lagkadinou E, Jia S, Pan H, Peng F, Ma Z, Wu Z, Guo X, Shi Y, Muik A, Sahin U, Zhu L, Zhu F. Safety and immunogenicity of the SARS-CoV-2 BNT162b1 mRNA vaccine in younger and older Chinese adults: a randomized, placebo-controlled, double-blind phase 1 study. Nat Med. 2021 Jun;27(6):1062-1070. doi: 10.1038/s41591-021-01330-9. Epub 2021 Apr 22. PMID 33888900
- [Background] Muik A, Lui BG, Wallisch AK, Bacher M, Muhl J, Reinholz J, Ozhelvaci O, Beckmann N, Guimil Garcia RC, Poran A, Shpyro S, Finlayson A, Cai H, Yang Q, Swanson KA, Tureci O, Sahin U. Neutralization of SARS-CoV-2 Omicron by BNT162b2 mRNA vaccine-elicited human sera. Science. 2022 Feb 11;375(6581):678-680. doi: 10.1126/science.abn7591. Epub 2022 Jan 18. PMID 35040667
- [Background] Quandt J, Muik A, Salisch N, Lui BG, Lutz S, Kruger K, Wallisch AK, Adams-Quack P, Bacher M, Finlayson A, Ozhelvaci O, Vogler I, Grikscheit K, Hoehl S, Goetsch U, Ciesek S, Tureci O, Sahin U. Omicron BA.1 breakthrough infection drives cross-variant neutralization and memory B cell formation against conserved epitopes. Sci Immunol. 2022 Sep 16;7(75):eabq2427. doi: 10.1126/sciimmunol.abq2427. Epub 2022 Sep 16. PMID 35653438
- [Derived] Pather S, Charpentier N, van den Ouweland F, Rizzi R, Finlayson A, Salisch N, Muik A, Lindemann C, Khanim R, Abduljawad S, Smith ER, Gurwith M, Chen RT; Benefit-Risk Assessment of VAccines by TechnolOgy Working Group (BRAVATO; ex-V3SWG). A Brighton Collaboration standardized template with key considerations for a benefit-risk assessment for the Comirnaty COVID-19 mRNA vaccine. Vaccine. 2024 Sep 17;42(22):126165. doi: 10.1016/j.vaccine.2024.126165. Epub 2024 Aug 27. PMID 39197299
- [Derived] Muik A, Lui BG, Bacher M, Wallisch AK, Toker A, Finlayson A, Kruger K, Ozhelvaci O, Grikscheit K, Hoehl S, Ciesek S, Tureci O, Sahin U. Omicron BA.2 breakthrough infection enhances cross-neutralization of BA.2.12.1 and BA.4/BA.5. Sci Immunol. 2022 Nov 25;7(77):eade2283. doi: 10.1126/sciimmunol.ade2283. Epub 2022 Nov 18. PMID 36125366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were selected from the volunteer panel at the clinical CRO, volunteers who responded to either generic or study-specific advertisements in social media, or volunteers who contacted the clinical CRO via a web-based study participant recruitment portal. Study participants were selected from this pool of volunteers according to inclusion and exclusion criteria. The first participant was enrolled on 23 APR 2020.
Pre-assignment Details: All enrolled participants were allocated to treatment.
Groups:
- BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg: BNT162a1: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (Prime/Boost [P/B] regimen).
- BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg: BNT162a1: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen).
- BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg: BNT162a1: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (Prime regimen only, as decided by the Safety Review Committee [SRC]).
- BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg; BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg; BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg; BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg; BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg; BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg; BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg; BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg; BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg: BNT162b1: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen).
- BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg: BNT162b1: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (Prime regimen only, as decided by the SRC).
- BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg; BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg; BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg; BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg; BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg; BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg; BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg; BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg: BNT162b2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen).
- BNT162b2 - Part A Immunocompromised (IC) Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13); BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13): BNT162b2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen), IC expansion cohort.
- BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11): BNT162b2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen), alternative posology dose group expansion cohort.
- BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12): BNT162b2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen), adaptive immune response dose group expansion cohort.
- BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14): BNT162b2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen), B-cell immune response dose group expansion cohort.
- BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B); BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B); BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B); BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B): BNT162c2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen).
- BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg Single Dose (SD); BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD); BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD); BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD): BNT162c2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (SD regimen).
Period: Overall Study
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Immunocompromised (IC) Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg Single Dose (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD)
Started | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 90 | 20 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed End of Treatment | 12 | 12 | 6 | 12 | 12 | 11 | 10 | 11 | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 89 | 19 | 12 | 12 | 12 | 11 | 12 | 12 | 11 | 12
Completed End of Follow-up Phase | 12 | 12 | 6 | 12 | 12 | 11 | 10 | 11 | 11 | 11 | 12 | 11 | 12 | 11 | 12 | 11 | 11 | 12 | 12 | 11 | 11 | 0 | 0 | 0 | 0 | 19 | 12 | 12 | 12 | 10 | 12 | 12 | 11 | 11
Completed | 12 | 12 | 6 | 12 | 12 | 11 | 10 | 11 | 11 | 11 | 12 | 11 | 12 | 11 | 12 | 11 | 11 | 12 | 12 | 11 | 11 | 0 | 0 | 0 | 0 | 19 | 12 | 12 | 12 | 10 | 12 | 12 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 15 | 15 | 30 | 90 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Private reason(s) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Roll-over into trial BNT162-14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11 | 10 | 31 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — non-trial SARS-COV-2 vaccination due to COVID-19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 16 | 55 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg; BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg: BNT162a1: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen).
- BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg: BNT162a1: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (Prime regimen only as decided by SRC).
- BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg: BNT162b1: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (Prime regimen only as decided by SRC).
- BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13); BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13): BNT162b2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen), IC expansion cohort.
- BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD); BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD); BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD); BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD): BNT162c2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (SD regimen).
- Total: Total of all reporting groups
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD) | Total
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 90 | 20 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 512
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.80 (2.58) | 48.31 (9.04) | 38.22 (13.87) | 38.21 (10.48) | 41.44 (11.27) | 43.62 (11.03) | 39.42 (11.41) | 35.74 (8.60) | 33.88 (10.72) | 35.81 (12.50) | 64.31 (5.89) | 65.66 (5.95) | 67.16 (6.47) | 36.65 (10.14) | 39.64 (10.14) | 35.07 (10.46) | 42.75 (9.89) | 47.21 (6.43) | 65.44 (7.42) | 65.88 (6.56) | 63.87 (5.42) | 48.04 (10.36) | 48.93 (11.87) | 51.92 (13.57) | 55.59 (16.07) | 48.45 (13.87) | 36.42 (10.33) | 39.41 (12.34) | 34.47 (10.24) | 35.42 (9.68) | 40.03 (14.67) | 35.23 (11.88) | 42.40 (12.04) | 32.60 (10.87) | 47.00 (15.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 1 | 7 | 6 | 8 | 4 | 4 | 6 | 5 | 5 | 10 | 8 | 5 | 7 | 8 | 10 | 4 | 4 | 6 | 8 | 3 | 9 | 13 | 45 | 10 | 8 | 5 | 3 | 8 | 10 | 8 | 5 | 7 | 261
  Male | 7 | 6 | 5 | 5 | 6 | 4 | 8 | 8 | 6 | 7 | 7 | 2 | 4 | 7 | 5 | 4 | 2 | 8 | 8 | 6 | 4 | 12 | 6 | 17 | 45 | 10 | 4 | 7 | 9 | 4 | 2 | 4 | 7 | 5 | 251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 6
  Not Hispanic or Latino | 12 | 12 | 6 | 11 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 89 | 20 | 12 | 12 | 10 | 12 | 12 | 11 | 12 | 12 | 506
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 12 | 12 | 5 | 12 | 12 | 11 | 11 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 14 | 15 | 30 | 89 | 19 | 11 | 11 | 12 | 12 | 12 | 11 | 12 | 12 | 502
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Germany | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 90 | 20 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 512
Weight [Mean (Standard Deviation); unit: kg] | 77.68 (7.59) | 72.54 (10.85) | 78.58 (14.93) | 72.99 (14.79) | 77.11 (14.07) | 71.57 (14.09) | 73.58 (11.88) | 79.84 (13.81) | 76.73 (13.32) | 78.70 (13.85) | 71.90 (10.98) | 70.38 (9.14) | 69.98 (8.06) | 80.18 (14.13) | 77.08 (10.84) | 76.11 (11.67) | 72.45 (10.97) | 77.78 (8.43) | 77.87 (9.78) | 76.91 (12.38) | 75.80 (11.98) | 73.85 (9.67) | 73.50 (10.07) | 77.79 (12.92) | 75.44 (13.02) | 79.09 (14.94) | 67.45 (13.53) | 76.41 (15.66) | 72.44 (6.86) | 70.94 (11.43) | 63.75 (6.14) | 73.26 (15.39) | 73.48 (9.51) | 68.90 (11.56) | 74.75 (12.27)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.61 (3.14) | 24.23 (2.78) | 24.73 (2.63) | 25.17 (2.89) | 24.94 (2.68) | 24.20 (2.32) | 24.34 (2.33) | 25.68 (3.44) | 25.52 (3.50) | 25.19 (3.09) | 24.73 (2.46) | 25.59 (2.22) | 25.63 (2.22) | 25.25 (3.26) | 25.50 (2.79) | 25.13 (2.07) | 25.43 (2.34) | 25.01 (1.38) | 25.43 (2.15) | 25.62 (2.47) | 25.85 (2.75) | 23.62 (1.90) | 25.63 (2.82) | 25.53 (2.72) | 25.08 (2.73) | 26.12 (2.96) | 23.31 (2.38) | 25.02 (2.85) | 23.83 (2.39) | 25.06 (3.73) | 22.82 (1.54) | 24.97 (3.17) | 24.19 (2.04) | 24.04 (2.59) | 24.98 (2.69)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Reactions at the Injection Site (Pain, Tenderness, Erythema/Redness, Induration/Swelling) Recorded up to 7 Days After Each IMP Dose.
Description: Solicited local reactions at the injection site (pain, tenderness, erythema/redness, and induration/swelling) were monitored and graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". The reporting of local reactions was based on the participant's assessments via daily solicited reports in the participant diaries.
Time Frame: From Day 1 to Day 8 for Dose 1 (Prime Immunization) and from Day 22 to Day 29 for Dose 2 (Boost Immunization)
Population: Safety Set - All subjects who received at least one dose of the IMP.
Measure: Count of Participants; unit: Participants
Groups:
- BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg: BNT162a1: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (Prime regimen only, as decided by the SRC).
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD)
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 90 | 20 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Participants
  Prime up to Day 7 after Prime: Number of participants with any local reaction | 9 | 11 | 6 | 6 | 5 | 10 | 12 | 11 | 12 | 12 | 7 | 11 | 11 | 6 | 9 | 12 | 12 | 10 | 7 | 9 | 9 | 12 | 14 | 16 | 82 | 20 | 4 | 3 | 8 | 11 | 4 | 7 | 5 | 11
  Prime up to Day 7 after Prime: Number of participants with any severe/grade >= 3 local reaction | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Boost up to Day 7 after Boost: Number of participants with any local reaction: number analyzed (Participants) | 12 | 12 | 0 | 12 | 12 | 11 | 11 | 12 | 11 | 0 | 12 | 11 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 89 | 19 | 12 | 12 | 12 | 11 | 0 | 0 | 0 | 0
  Boost up to Day 7 after Boost: Number of participants with any local reaction | 3 | 10 |  | 7 | 5 | 10 | 11 | 11 | 11 |  | 8 | 9 | 9 | 4 | 8 | 10 | 10 | 11 | 7 | 8 | 10 | 12 | 11 | 27 | 79 | 19 | 3 | 5 | 7 | 8 |  |  |  |
  Boost up to Day 7 after Boost: Number of participants with any severe/grade >= 3 local reaction: number analyzed (Participants) | 12 | 12 | 0 | 12 | 12 | 11 | 11 | 12 | 11 | 0 | 12 | 11 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 89 | 19 | 12 | 12 | 12 | 11 | 0 | 0 | 0 | 0
  Boost up to Day 7 after Boost: Number of participants with any severe/grade >= 3 local reaction | 0 | 0 |  | 2 | 0 | 0 | 0 | 2 | 3 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 |  |  |  |

2. Primary Outcome: Number of Participants With Solicited Systemic Reactions (Nausea, Vomiting, Diarrhea, Headache, Fatigue, Myalgia, Arthralgia, Chills, Loss of Appetite, Malaise, and Fever) Recorded up to 7 Days After Each IMP Dose.
Description: Solicited systemic reactions (nausea, vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills, loss of appetite, malaise, and fever) were monitored and graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". The reporting of systemic reactions was based on the participant's assessments via daily solicited reports in the participant diaries.
Time Frame: From Day 1 to Day 8 for Dose 1 (Prime Immunization) and from Day 22 to Day 29 for Dose 2 (Boost Immunization)
Population: Safety Set - All subjects who received at least one dose of the IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD)
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 90 | 20 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Participants
  Prime up to Day 7 after Prime: Number of participants with any systemic reaction | 6 | 12 | 6 | 9 | 8 | 8 | 11 | 11 | 12 | 12 | 9 | 10 | 11 | 9 | 9 | 12 | 9 | 9 | 3 | 4 | 9 | 12 | 14 | 12 | 68 | 15 | 5 | 8 | 9 | 12 | 7 | 7 | 4 | 8
  Prime up to Day 7 after Prime: Number of participants with any severe / grade >= 3 systemic reaction | 1 | 1 | 5 | 0 | 0 | 1 | 2 | 3 | 5 | 8 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2
  Boost up to Day 7 after Boost: Number of participants with any systemic reaction: number analyzed (Participants) | 12 | 12 | 0 | 12 | 12 | 11 | 11 | 12 | 11 | 0 | 12 | 11 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 89 | 19 | 12 | 12 | 12 | 11 | 0 | 0 | 0 | 0
  Boost up to Day 7 after Boost: Number of participants with any systemic reaction | 3 | 12 |  | 7 | 7 | 9 | 10 | 11 | 11 |  | 8 | 10 | 12 | 4 | 2 | 7 | 10 | 10 | 4 | 8 | 11 | 13 | 12 | 21 | 78 | 16 | 3 | 7 | 6 | 9 |  |  |  |
  Boost up to Day 7 after Boost: Number of participants with any severe / grade >= 3 systemic reaction: number analyzed (Participants) | 12 | 12 | 0 | 12 | 12 | 11 | 11 | 12 | 11 | 0 | 12 | 11 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 89 | 19 | 12 | 12 | 12 | 11 | 0 | 0 | 0 | 0
  Boost up to Day 7 after Boost: Number of participants with any severe / grade >= 3 systemic reaction | 0 | 4 |  | 3 | 1 | 5 | 5 | 6 | 5 |  | 2 | 2 | 4 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 2 | 4 | 1 | 4 | 14 | 3 | 1 | 1 | 0 | 2 |  |  |  |

3. Primary Outcome: The Percentage of Participants With at Least 1 Unsolicited Treatment Emergent Adverse Event (TEAE) Occurring After Dose 1 (Prime Immunization) up to Dose 2 (Boost Immunization) or 28 Days After Dose 1.
Description: TEAEs without AEs based on solicited reporting via diaries, were analyzed by vaccine, age group, dose level, and for each IMP dose. The percentage of participants reporting at least one TEAE was summarized by adverse event types (any TEAE and any grade >=3 TEAE) using the Safety Set.
Time Frame: 28 days following Dose 1 or up to Dose 2 (whichever was first)
Population: Safety Set - All participants who received at least one dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD)
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 90 | 20 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
percentage of participants
  Any TEAE | 8 | 33 | 83 | 8 | 0 | 50 | 33 | 42 | 42 | 58 | 25 | 17 | 58 | 25 | 50 | 50 | 8 | 42 | 25 | 33 | 25 | 7 | 53 | 13 | 26 | 35 | 17 | 33 | 17 | 17 | 50 | 58 | 25 | 25
  Any grade >=3 TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 8 | 8 | 8 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 17 | 0 | 7 | 0 | 2 | 5 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0

4. Primary Outcome: The Percentage of Participants With at Least 1 Unsolicited TEAE Occurring After Dose 1 up to 28 Days After Dose 2 (Boost Immunization) or After Dose 1 (Prime Immunization) (if no Dose 2)
Description: TEAEs, without AEs based on solicited reporting via diaries, were analyzed by vaccine, age group, dose level, and for each IMP dose. The percentage of participants reporting at least one TEAE was summarized by adverse event types (any TEAE and any grade >=3 TEAE) using the Safety Set.
Time Frame: 28 days following Dose 2 or Dose 1 (if no Dose 2 was given)
Population: Safety Set - All participants who received at least one dose of the IMP. Per study protocol, this endpoint was only applicable for arms planned to receive two doses.
Measure: Number; unit: percentage of participants
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B)
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 15 | 15 | 30 | 90 | 20 | 12 | 12 | 12 | 12
percentage of participants
  Any TEAE | 17 | 33 | 83 | 58 | 8 | 75 | 50 | 58 | 67 | 58 | 25 | 33 | 75 | 58 | 58 | 67 | 25 | 50 | 33 | 58 | 33 | 13 | 73 | 40 | 49 | 45 | 33 | 42 | 33 | 17
  Any grade >=3 TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 0 | 0 | 0 | 8 | 8 | 17 | 0 | 0 | 8 | 0 | 0 | 8 | 8 | 17 | 0 | 7 | 3 | 4 | 10 | 0 | 8 | 0 | 8

5. Secondary Outcome: Functional Antibody Responses (Titers) for BNT162a1, BNT162b1, BNT162b2 (Younger and Older Dose Ranging Cohorts), and BNT162c2 (P/B)
Description: At Day 1 (Baseline = Pre-Prime Immunization) and at 7 and 21 days after Dose 1 (Prime Immunization) and at 7, 21, 28, 63, and 162 days after Dose 2 (Boost Immunization).
Time Frame: up to 183 days following Dose 1
Population: Immunogenicity set - all participants who received at least one dose of IMP and had at least one post-baseline functional antibody titer immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B)
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
titer
  Day 1 (Baseline = Pre-Prime Immunization) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.1 [4.8 to 5.5] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 6.9 [3.4 to 13.8] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  7 days after Dose 1 (Day 8): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 11
  7 days after Dose 1 (Day 8) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.1 [4.8 to 5.5] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 8.2 [2.8 to 24.1] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  21 days after Dose 1 (Day 22): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
  21 days after Dose 1 (Day 22) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 10.0 [6.1 to 16.3] | 6.9 [4.4 to 10.7] | 10.0 [5.4 to 18.5] | 11.7 [6.2 to 22.1] | 29.1 [13.5 to 63.0] | 20.6 [11.5 to 37.0] | 13.7 [7.5 to 25.3] | 16.3 [7.7 to 34.5] | 15.4 [7.8 to 30.4] | 16.3 [8.3 to 32.3] | 5.3 [4.7 to 6.0] | 7.5 [5.6 to 10.1] | 16.6 [9.7 to 28.3] | 16.3 [8.0 to 33.5] | 15.9 [9.6 to 26.2] | 8.4 [5.6 to 12.6] | 7.9 [5.2 to 12.1] | 49.0 [18.3 to 131.4] | 5.0 [5.0 to 5.0] | 5.3 [4.7 to 6.0] | 5.3 [4.7 to 6.0] | 7.1 [4.9 to 10.2]
  7 days after Dose 2 (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 0 | 11 | 0 | 0 | 0 | 12 | 12 | 12 | 12 | 12 | 1 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 11
  7 days after Dose 2 (Day 29) |  |  |  |  | 55.0 [32.5 to 93.1] |  | 181.5 [107.5 to 306.3] |  |  |  | 320.0 [183.6 to 557.7] | 169.5 [70.3 to 408.7] | 207.5 [94.0 to 458.0] | 38.9 [16.1 to 93.5] | 134.5 [82.2 to 220.1] | 40.0 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available. | 213.6 [114.7 to 397.7] | 329.4 [203.2 to 533.9] | 127.0 [79.2 to 203.7] | 164.7 [77.0 to 352.0] | 678.1 [395.9 to 1161.2] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.3 [4.7 to 6.0] | 8.0 [4.8 to 13.4]
  21 days after Dose 2 (Day 43): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 10 | 12 | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 11 | 11
  21 days after Dose 2 (Day 43) | 5.0 [5.0 to 5.0] | 8.7 [3.8 to 19.8] | 5.3 [4.6 to 6.1] | 69.2 [33.0 to 145.4] | 95.1 [47.0 to 192.7] | 62.2 [30.4 to 127.0] | 160.0 [90.3 to 283.6] | 184.9 [96.8 to 353.0] | 282.1 [136.8 to 581.6] | 8.9 [6.1 to 13.0] | 293.4 [179.9 to 478.5] | 95.1 [42.3 to 214.0] | 134.5 [66.8 to 270.8] | 49.9 [26.9 to 92.6] | 109.9 [71.1 to 169.8] | 187.3 [119.9 to 292.6] | 164.7 [89.3 to 303.6] | 300.5 [182.7 to 494.1] | 134.5 [84.5 to 214.1] | 169.5 [115.3 to 249.2] | 452.5 [255.6 to 801.1] | 5.1 [4.8 to 5.5] | 5.6 [4.9 to 6.5] | 5.7 [4.8 to 6.6] | 6.0 [4.6 to 8.0]
  28 days after Dose 2 (Day 50): number analyzed (Participants) | 2 | 0 | 0 | 0 | 12 | 0 | 12 | 0 | 0 | 0 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12
  28 days after Dose 2 (Day 50) | 5.0 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available. |  |  |  | 80.0 [36.1 to 177.5] |  | 82.3 [37.4 to 181.1] |  |  |  | 226.3 [120.5 to 424.8] | 89.8 [37.5 to 214.9] | 95.1 [50.9 to 178.0] | 36.4 [20.8 to 63.8] | 67.3 [35.7 to 126.7] | 190.3 [118.4 to 305.7] | 160.0 [84.6 to 302.5] | 213.6 [148.8 to 306.6] | 127.0 [75.7 to 213.0] | 132.4 [91.8 to 191.0] | 391.7 [229.4 to 668.8] | 5.0 [5.0 to 5.0] | 5.9 [5.0 to 7.1] | 5.0 [5.0 to 5.0] | 5.3 [4.7 to 6.0]
  63 days after Dose 2 (Day 85): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 10 | 11 | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 11 | 12 | 12 | 11 | 12 | 8
  63 days after Dose 2 (Day 85) | 5.0 [5.0 to 5.0] | 7.5 [3.9 to 14.5] | 5.0 [5.0 to 5.0] | 25.9 [14.6 to 46.0] | 31.7 [14.5 to 69.4] | 40.0 [21.1 to 76.0] | 134.5 [70.0 to 258.6] | 102.9 [58.1 to 182.2] | 120.5 [56.1 to 258.7] | 7.7 [5.2 to 11.4] | 46.2 [25.4 to 84.0] | 33.6 [16.6 to 68.1] | 69.2 [33.8 to 142.0] | 36.4 [19.3 to 68.6] | 33.6 [19.9 to 57.0] | 145.6 [85.5 to 247.8] | 146.7 [80.9 to 265.9] | 160.0 [97.4 to 263.0] | 21.8 [12.1 to 39.2] | 27.4 [17.5 to 42.9] | 80.0 [39.1 to 163.5] | 5.6 [5.0 to 6.3] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.2 [4.7 to 5.8]
  162 days after Dose 2 (Day 184): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 11 | 11 | 11 | 11 | 12 | 11 | 12 | 11 | 12 | 11 | 11 | 12 | 12 | 11 | 11 | 12 | 12 | 12 | 10
  162 days after Dose 2 (Day 184) | 5.0 [5.0 to 5.0] | 6.9 [3.4 to 13.8] | 5.0 [5.0 to 5.0] | 10.0 [6.1 to 16.4] | 15.0 [9.0 to 24.8] | 13.7 [8.8 to 21.4] | 27.4 [14.0 to 53.6] | 29.2 [13.9 to 61.2] | 56.6 [22.3 to 143.6] | 5.2 [4.8 to 5.5] | 16.8 [10.0 to 28.2] | 19.4 [10.7 to 35.1] | 65.4 [31.7 to 134.8] | 8.5 [5.6 to 13.0] | 11.2 [7.8 to 16.2] | 21.3 [12.2 to 37.3] | 54.8 [31.5 to 95.5] | 38.9 [20.6 to 73.2] | 26.7 [14.1 to 50.4] | 15.5 [11.8 to 20.5] | 58.4 [30.6 to 111.3] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.8 [4.2 to 7.9] | 10.4 [3.4 to 31.5]

6. Secondary Outcome: Fold Increase in Functional Antibody Titers as Compared to Baseline for BNT162a1, BNT162b1, BNT162b2 (Younger and Older Dose Ranging Cohorts), and BNT162c2 (P/B)
Description: At 7 and 21 days after Dose 1 (Prime Immunization) and at 7, 21, 28, 63, and 162 days after Dose 2 (Boost Immunization).
Time Frame: up to 183 days following Dose 1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B)
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Fold rise
  7 days after Dose 1 (Day 8): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 11
  7 days after Dose 1 (Day 8) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.2 [0.8 to 1.7] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  21 days after Dose 1 (Day 22): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
  21 days after Dose 1 (Day 22) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 2.0 [1.2 to 3.3] | 1.4 [0.9 to 2.1] | 2.0 [1.1 to 3.7] | 2.3 [1.2 to 4.4] | 5.8 [2.7 to 12.6] | 4.0 [2.2 to 7.3] | 2.7 [1.5 to 5.1] | 3.3 [1.5 to 6.9] | 3.1 [1.6 to 6.1] | 3.3 [1.7 to 6.5] | 1.1 [0.9 to 1.2] | 1.5 [1.1 to 2.0] | 3.3 [1.9 to 5.7] | 3.3 [1.6 to 6.7] | 3.2 [1.9 to 5.2] | 1.7 [1.1 to 2.5] | 1.6 [1.0 to 2.4] | 7.1 [4.3 to 11.9] | 1.0 [1.0 to 1.0] | 1.1 [0.9 to 1.2] | 1.1 [0.9 to 1.2] | 1.4 [1.0 to 2.0]
  7 days after Dose 2 (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 0 | 11 | 0 | 0 | 0 | 12 | 12 | 12 | 12 | 12 | 1 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 11
  7 days after Dose 2 (Day 29) |  |  |  |  | 11.0 [6.5 to 18.6] |  | 36.3 [21.5 to 61.3] |  |  |  | 64.0 [36.7 to 111.5] | 33.9 [14.1 to 81.7] | 41.5 [18.8 to 91.6] | 7.8 [3.2 to 18.7] | 26.9 [16.4 to 44.0] | 8.0 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available. | 42.7 [22.9 to 79.5] | 65.9 [40.6 to 106.8] | 25.4 [15.8 to 40.7] | 32.9 [15.4 to 70.4] | 98.7 [62.2 to 156.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.1 [0.9 to 1.2] | 1.6 [1.0 to 2.7]
  21 days after Dose 2 (Day 43): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 10 | 12 | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 11 | 11
  21 days after Dose 2 (Day 43) | 1.0 [1.0 to 1.0] | 1.7 [0.8 to 4.0] | 1.1 [0.9 to 1.2] | 13.8 [6.6 to 29.1] | 19.0 [9.4 to 38.5] | 12.4 [6.1 to 25.4] | 32.0 [18.1 to 56.7] | 37.0 [19.4 to 70.6] | 54.7 [26.5 to 112.8] | 1.8 [1.2 to 2.6] | 58.7 [36.0 to 95.7] | 19.0 [8.5 to 42.8] | 26.9 [13.4 to 54.2] | 10.0 [5.4 to 18.5] | 22.0 [14.2 to 34.0] | 37.5 [24.0 to 58.5] | 32.9 [17.9 to 60.7] | 60.1 [36.5 to 98.8] | 26.9 [16.9 to 42.8] | 33.9 [23.1 to 49.8] | 65.9 [45.5 to 95.3] | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.3] | 1.1 [1.0 to 1.3] | 1.2 [0.9 to 1.6]
  28 days after Dose 2 (Day 50): number analyzed (Participants) | 2 | 0 | 0 | 0 | 12 | 0 | 12 | 0 | 0 | 0 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12
  28 days after Dose 2 (Day 50) | 1.0 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available. |  |  |  | 16.0 [7.2 to 35.5] |  | 16.5 [7.5 to 36.2] |  |  |  | 45.3 [24.1 to 85.0] | 18.0 [7.5 to 43.0] | 19.0 [10.2 to 35.6] | 7.3 [4.2 to 12.8] | 13.5 [7.1 to 25.3] | 38.1 [23.7 to 61.1] | 32.0 [16.9 to 60.5] | 42.7 [29.8 to 61.3] | 25.4 [15.1 to 42.6] | 26.5 [18.4 to 38.2] | 57.0 [38.6 to 84.3] | 1.0 [1.0 to 1.0] | 1.2 [1.0 to 1.4] | 1.0 [1.0 to 1.0] | 1.1 [0.9 to 1.2]
  63 days after Dose 2 (Day 85): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 10 | 11 | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 11 | 12 | 12 | 11 | 12 | 8
  63 days after Dose 2 (Day 85) | 1.0 [1.0 to 1.0] | 1.5 [0.8 to 2.9] | 1.0 [1.0 to 1.0] | 5.2 [2.9 to 9.2] | 6.3 [2.9 to 13.9] | 8.0 [4.2 to 15.2] | 26.9 [14.0 to 51.7] | 20.6 [11.6 to 36.4] | 23.4 [10.8 to 50.4] | 1.5 [1.0 to 2.3] | 9.2 [5.1 to 16.8] | 6.7 [3.3 to 13.6] | 13.8 [6.8 to 28.4] | 7.3 [3.9 to 13.7] | 6.7 [4.0 to 11.4] | 29.1 [17.1 to 49.6] | 29.3 [16.2 to 53.2] | 32.0 [19.5 to 52.6] | 4.4 [2.4 to 7.8] | 5.5 [3.5 to 8.6] | 11.6 [7.3 to 18.7] | 1.1 [1.0 to 1.3] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [0.9 to 1.2]
  162 days after Dose 2 (Day 184): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 11 | 11 | 11 | 11 | 12 | 11 | 12 | 11 | 12 | 11 | 11 | 12 | 12 | 11 | 11 | 12 | 12 | 12 | 10
  162 days after Dose 2 (Day 184) | 1.0 [1.0 to 1.0] | 1.4 [0.7 to 2.8] | 1.0 [1.0 to 1.0] | 2.0 [1.2 to 3.3] | 3.0 [1.8 to 5.0] | 2.7 [1.8 to 4.3] | 5.5 [2.8 to 10.7] | 5.8 [2.8 to 12.2] | 11.0 [4.3 to 28.2] | 1.0 [1.0 to 1.1] | 3.4 [2.0 to 5.6] | 3.9 [2.1 to 7.0] | 13.1 [6.3 to 27.0] | 1.7 [1.1 to 2.6] | 2.2 [1.6 to 3.2] | 4.3 [2.4 to 7.5] | 11.0 [6.3 to 19.1] | 7.8 [4.1 to 14.6] | 5.3 [2.8 to 10.1] | 3.1 [2.4 to 4.1] | 11.7 [6.1 to 22.3] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.2 [0.8 to 1.6] | 2.1 [0.7 to 6.3]

7. Secondary Outcome: Number of Participants With Seroconversion Defined as a Minimum of 4-fold Increase of Functional Antibody Titers as Compared to Baseline for BNT162a1, BNT162b1, BNT162b2 (Younger and Older Dose Ranging Cohorts), and BNT162c2 (P/B)
Description: At 7 and 21 days after Dose 1 (Prime Immunization) and at 7, 21, 28, 63, and 162 days after Dose 2 (Boost Immunization).
Time Frame: up to 183 days following Dose 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B)
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Participants
  7 days after Dose 1 (Day 8): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 11
  7 days after Dose 1 (Day 8) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  21 days after Dose 1 (Day 22): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
  21 days after Dose 1 (Day 22) | 0 | 0 | 0 | 2 | 1 | 3 | 3 | 7 | 7 | 6 | 5 | 6 | 3 | 0 | 0 | 7 | 5 | 6 | 2 | 2 | 10 | 0 | 0 | 0 | 1
  7 days after Dose 2 (Day 29): number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 0 | 11 | 0 | 0 | 0 | 12 | 12 | 12 | 12 | 12 | 1 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 11
  7 days after Dose 2 (Day 29) |  |  |  |  | 11 |  | 11 |  |  |  | 12 | 12 | 11 | 7 | 12 | 1 | 12 | 12 | 12 | 12 | 12 | 0 | 0 | 0 | 2
  21 days after Dose 2 (Day 43): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 10 | 12 | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 11 | 11
  21 days after Dose 2 (Day 43) | 0 | 2 | 0 | 10 | 11 | 9 | 10 | 12 | 11 | 3 | 12 | 11 | 12 | 9 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 0 | 0 | 0 | 0
  28 days after Dose 2 (Day 50): number analyzed (Participants) | 2 | 0 | 0 | 0 | 12 | 0 | 12 | 0 | 0 | 0 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 12 | 12 | 12 | 12
  28 days after Dose 2 (Day 50) | 0 |  |  |  | 11 |  | 11 |  |  |  | 12 | 11 | 12 | 9 | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 0 | 0 | 0 | 0
  63 days after Dose 2 (Day 85): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 10 | 11 | 11 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12 | 12 | 12 | 11 | 12 | 12 | 11 | 12 | 8
  63 days after Dose 2 (Day 85) | 0 | 2 | 0 | 9 | 8 | 9 | 10 | 11 | 11 | 1 | 10 | 8 | 10 | 8 | 9 | 11 | 12 | 12 | 8 | 7 | 12 | 0 | 0 | 0 | 0
  162 days after Dose 2 (Day 184): number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 11 | 11 | 11 | 11 | 11 | 12 | 11 | 12 | 11 | 12 | 11 | 11 | 12 | 12 | 11 | 11 | 12 | 12 | 12 | 10
  162 days after Dose 2 (Day 184) | 0 | 1 | 0 | 3 | 6 | 4 | 7 | 8 | 10 | 0 | 5 | 7 | 10 | 3 | 2 | 6 | 10 | 11 | 7 | 4 | 10 | 0 | 0 | 1 | 2

8. Secondary Outcome: Functional Antibody Responses (Titers) for BNT162c2 (SD)
Description: At Day 1 (Baseline = Pre Immunization) and at 7, 21, 28, 42, 84, and 183 days after Dose 1 (Prime Immunization).
Time Frame: up to 183 days following Dose 1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD)
Number analyzed (Participants) | 12 | 12 | 12 | 12
titer
  Day 1 (Baseline = Pre Immunization) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  7 days after Dose 1 (Day 8) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  21 days after Dose 1 (Day 22) | 5.1 [4.8 to 5.5] | 5.1 [4.8 to 5.5] | 5.3 [4.7 to 6.0] | 5.5 [4.8 to 6.3]
  28 days after Dose 1 (Day 29): number analyzed (Participants) | 0 | 12 | 9 | 10
  28 days after Dose 1 (Day 29) |  | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.2 [4.8 to 5.6]
  42 days after Dose 1 (Day 43) | 5.1 [4.8 to 5.5] | 5.1 [4.8 to 5.5] | 5.5 [4.5 to 6.6] | 5.1 [4.8 to 5.5]
  84 days after Dose 1 (Day 85): number analyzed (Participants) | 11 | 12 | 11 | 11
  84 days after Dose 1 (Day 85) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 6.0 [4.0 to 9.2] | 5.0 [5.0 to 5.0]
  183 days after Dose 1 (Day 184): number analyzed (Participants) | 12 | 12 | 11 | 11
  183 days after Dose 1 (Day 184) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.5 [4.5 to 6.8] | 6.4 [3.7 to 11.3]

9. Secondary Outcome: Fold Increase in Functional Antibody Titers as Compared to Baseline for BNT162c2 (SD)
Description: At 7, 21, 28, 42, 84, and 183 days after Dose 1 (Prime Immunization).
Time Frame: up to 183 days following Dose 1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Fold rise
  7 days after Dose 1 (Day 8) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  21 days after Dose 1 (Day 22) | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.1 [0.9 to 1.2] | 1.1 [1.0 to 1.3]
  28 days after Dose 1 (Day 29): number analyzed (Participants) | 0 | 12 | 9 | 10
  28 days after Dose 1 (Day 29) |  | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1]
  42 days after Dose 1 (Day 43) | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.1 [0.9 to 1.3] | 1.0 [1.0 to 1.1]
  84 days after Dose 1 (Day 85): number analyzed (Participants) | 11 | 12 | 11 | 11
  84 days after Dose 1 (Day 85) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.2 [0.8 to 1.8] | 1.0 [1.0 to 1.0]
  183 days after Dose 1 (Day 184): number analyzed (Participants) | 12 | 12 | 11 | 11
  183 days after Dose 1 (Day 184) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.1 [0.9 to 1.4] | 1.3 [0.7 to 2.3]

10. Secondary Outcome: Number of Participants With Seroconversion Defined as a Minimum of 4-fold Increase of Functional Antibody Titers as Compared to Baseline for BNT162c2 (SD)
Description: At 7, 21, 28, 42, 84, and 183 days after Dose 1 (Prime Immunization).
Time Frame: up to 183 days following Dose 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  7 days after Dose 1 (Day 8) | 0 | 0 | 0 | 0
  21 days after Dose 1 (Day 22) | 0 | 0 | 0 | 0
  28 days after Dose 1 (Day 29): number analyzed (Participants) | 0 | 12 | 9 | 10
  28 days after Dose 1 (Day 29) |  | 0 | 0 | 0
  42 days after Dose 1 (Day 43) | 0 | 0 | 0 | 0
  84 days after Dose 1 (Day 85): number analyzed (Participants) | 11 | 12 | 11 | 11
  84 days after Dose 1 (Day 85) | 0 | 0 | 1 | 0
  183 days after Dose 1 (Day 184): number analyzed (Participants) | 12 | 12 | 11 | 11
  183 days after Dose 1 (Day 184) | 0 | 0 | 0 | 1

11. Secondary Outcome: Functional Antibody Responses (Titers) for BNT162b2 (Expansion Cohorts 11, 12, 13, and 14; P/B)
Description: At Day 1 (Baseline = Pre-Prime Immunization) and at 7, 14, and 21 days after Dose 1 (Prime Immunization) and at 7, 14, 21, 28, 63, 162, and 343 days after Dose 2 (Boost Immunization).
Time Frame: up to 1 year following Dose 1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14)
Number analyzed (Participants) | 15 | 15 | 30 | 90 | 20
Titer
  Day 1 (Baseline = Pre-Prime Immunization) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.1 [4.9 to 5.3] | 5.0 [5.0 to 5.0]
  7 days after Dose 1 (Day 8) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.4 [4.8 to 6.0] | 5.3 [4.7 to 6.1] | 6.6 [4.2 to 10.4]
  14 days after Dose 1 (Day 15): number analyzed (Participants) | 0 | 0 | 0 | 0 | 20
  14 days after Dose 1 (Day 15) |  |  |  |  | 9.5 [4.8 to 18.7]
  21 days after Dose 1 (Day 22): number analyzed (Participants) | 15 | 15 | 30 | 89 | 19
  21 days after Dose 1 (Day 22) | 17.4 [9.8 to 30.9] | 5.2 [4.7 to 5.8] | 5.7 [4.8 to 6.8] | 21.9 [17.5 to 27.3] | 17.9 [9.5 to 33.7]
  7 days after Dose 2 (Day 29): number analyzed (Participants) | 15 | 15 | 30 | 89 | 19
  7 days after Dose 2 (Day 29) | 167.6 [112.0 to 250.7] | 12.0 [5.5 to 26.4] | 30.7 [21.3 to 44.1] | 348.6 [270.8 to 448.8] | 286.8 [183.1 to 449.4]
  14 days after Dose 2 (Day 36): number analyzed (Participants) | 15 | 15 | 30 | 88 | 0
  14 days after Dose 2 (Day 36) | 206.3 [116.8 to 364.3] | 11.5 [5.3 to 24.8] | 149.3 [104.0 to 214.4] | 379.1 [306.0 to 469.6] |
  21 days after Dose 2 (Day 43): number analyzed (Participants) | 15 | 15 | 30 | 89 | 0
  21 days after Dose 2 (Day 43) | 167.6 [93.8 to 299.2] | 9.8 [4.8 to 19.7] | 119.9 [81.5 to 176.4] | 307.8 [250.0 to 378.9] |
  28 days after Dose 2 (Day 50): number analyzed (Participants) | 15 | 15 | 30 | 89 | 19
  28 days after Dose 2 (Day 50) | 136.1 [76.2 to 243.0] | 11.0 [5.1 to 23.7] | 87.7 [62.3 to 123.7] | 266.5 [215.9 to 328.8] | 103.3 [70.8 to 150.6]
  63 days after Dose 2 (Day 85): number analyzed (Participants) | 15 | 15 | 30 | 89 | 0
  63 days after Dose 2 (Day 85) | 50.4 [30.7 to 82.7] | 8.3 [5.0 to 13.7] | 79.1 [56.7 to 110.2] | 99.9 [81.3 to 122.7] |
  162 days after Dose 2 (Day 184): number analyzed (Participants) | 15 | 12 | 24 | 89 | 19
  162 days after Dose 2 (Day 184) | 27.0 [16.3 to 44.6] | 11.9 [4.0 to 35.3] | 19.2 [11.9 to 30.9] | 29.5 [23.5 to 37.1] | 49.8 [33.3 to 74.4]
  343 days after Dose 2 (Day 365): number analyzed (Participants) | 0 | 0 | 1 | 16 | 0
  343 days after Dose 2 (Day 365) |  |  | 7.1 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available. | 30.2 [11.7 to 78.2] |

12. Secondary Outcome: Fold Increase in Functional Antibody Titers as Compared to Baseline for BNT162b2 (Expansion Cohorts 11, 12, 13, and 14; P/B)
Description: At 7, 14, and 21 days after Dose 1 (Prime Immunization) and at 7, 14, 21, 28, 63, 162, and 343 days after Dose 2 (Boost Immunization).
Time Frame: up to 1 year following Dose 1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14)
Number analyzed (Participants) | 15 | 15 | 30 | 90 | 20
Fold rise
  7 days after Dose 1 (Day 8) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.1] | 1.3 [0.8 to 2.1]
  14 days after Dose 1 (Day 15): number analyzed (Participants) | 0 | 0 | 0 | 0 | 20
  14 days after Dose 1 (Day 15) |  |  |  |  | 1.9 [1.0 to 3.7]
  21 days after Dose 1 (Day 22): number analyzed (Participants) | 15 | 15 | 30 | 89 | 19
  21 days after Dose 1 (Day 22) | 3.5 [2.0 to 6.2] | 1.0 [0.9 to 1.2] | 1.1 [1.0 to 1.4] | 4.3 [3.5 to 5.3] | 3.6 [1.9 to 6.7]
  7 days after Dose 2 (Day 29): number analyzed (Participants) | 15 | 15 | 30 | 89 | 19
  7 days after Dose 2 (Day 29) | 33.5 [22.4 to 50.1] | 2.4 [1.1 to 5.3] | 6.1 [4.3 to 8.8] | 68.4 [53.3 to 87.7] | 57.4 [36.6 to 89.9]
  14 days after Dose 2 (Day 36): number analyzed (Participants) | 15 | 15 | 30 | 88 | 0
  14 days after Dose 2 (Day 36) | 41.3 [23.4 to 72.9] | 2.3 [1.1 to 5.0] | 29.9 [20.8 to 42.9] | 74.3 [60.2 to 91.8] |
  21 days after Dose 2 (Day 43): number analyzed (Participants) | 15 | 15 | 30 | 89 | 0
  21 days after Dose 2 (Day 43) | 33.5 [18.8 to 59.8] | 2.0 [1.0 to 3.9] | 24.0 [16.3 to 35.3] | 60.4 [49.2 to 74.1] |
  28 days after Dose 2 (Day 50): number analyzed (Participants) | 15 | 15 | 30 | 89 | 19
  28 days after Dose 2 (Day 50) | 27.2 [15.2 to 48.6] | 2.2 [1.0 to 4.7] | 17.5 [12.5 to 24.7] | 52.3 [42.7 to 64.0] | 20.7 [14.2 to 30.1]
  63 days after Dose 2 (Day 85): number analyzed (Participants) | 15 | 15 | 30 | 89 | 0
  63 days after Dose 2 (Day 85) | 10.1 [6.1 to 16.5] | 1.7 [1.0 to 2.7] | 15.8 [11.3 to 22.0] | 19.6 [16.0 to 23.9] |
  162 days after Dose 2 (Day 184): number analyzed (Participants) | 15 | 12 | 24 | 89 | 19
  162 days after Dose 2 (Day 184) | 5.4 [3.3 to 8.9] | 2.4 [0.8 to 7.1] | 3.8 [2.4 to 6.2] | 5.8 [4.6 to 7.2] | 10.0 [6.7 to 14.9]
  343 days after Dose 2 (Day 365): number analyzed (Participants) | 0 | 0 | 1 | 16 | 0
  343 days after Dose 2 (Day 365) |  |  | 1.4 [NA to NA] — Confidence intervals were only calculated if values of at least 3 participants were available. | 5.4 [2.1 to 13.8] |

13. Secondary Outcome: Number of Participants With Seroconversion Defined as a Minimum of 4-fold Increase of Functional Antibody Titers as Compared to Baseline for BNT162b2 (Expansion Cohorts 11, 12, 13, and 14; P/B)
Description: as for outcome 12
Time Frame: up to 1 year following Dose 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14)
Number analyzed (Participants) | 15 | 15 | 30 | 90 | 20
Participants
  7 days after Dose 1 (Day 8) | 0 | 0 | 1 | 1 | 2
  14 days after Dose 1 (Day 15): number analyzed (Participants) | 0 | 0 | 0 | 0 | 20
  14 days after Dose 1 (Day 15) |  |  |  |  | 4
  21 days after Dose 1 (Day 22): number analyzed (Participants) | 15 | 15 | 30 | 89 | 19
  21 days after Dose 1 (Day 22) | 7 | 0 | 1 | 54 | 9
  7 days after Dose 2 (Day 29): number analyzed (Participants) | 15 | 15 | 30 | 89 | 19
  7 days after Dose 2 (Day 29) | 15 | 4 | 22 | 88 | 19
  14 days after Dose 2 (Day 36): number analyzed (Participants) | 15 | 15 | 30 | 88 | 0
  14 days after Dose 2 (Day 36) | 15 | 4 | 30 | 88 |
  21 days after Dose 2 (Day 43): number analyzed (Participants) | 15 | 15 | 30 | 89 | 0
  21 days after Dose 2 (Day 43) | 15 | 3 | 29 | 89 |
  28 days after Dose 2 (Day 50): number analyzed (Participants) | 15 | 15 | 30 | 89 | 19
  28 days after Dose 2 (Day 50) | 15 | 4 | 30 | 89 | 19
  63 days after Dose 2 (Day 85): number analyzed (Participants) | 15 | 15 | 30 | 89 | 0
  63 days after Dose 2 (Day 85) | 13 | 2 | 28 | 84 |
  162 days after Dose 2 (Day 184): number analyzed (Participants) | 15 | 12 | 24 | 89 | 19
  162 days after Dose 2 (Day 184) | 12 | 3 | 12 | 61 | 18
  343 days after Dose 2 (Day 365): number analyzed (Participants) | 0 | 0 | 1 | 16 | 0
  343 days after Dose 2 (Day 365) |  |  | 0 | 10 |

ADVERSE EVENTS:
Time Frame: Local reactions/systemic events: within 7 days after each IMP dose; SAEs: from Day 1 (Dose 1 [Prime Immunization]) up to Day 387 (approximately 12 months after Dose 2 [Boost Immunization]); Other AEs in participants with Dose 2: All AEs from Day 1 up to Day 50 and in addition if assessed as IMP-related from Day 50 up to Day 387; Other AEs in participants without Dose 2: All AEs from Day 1 up to Day 29 and in addition if assessed as IMP-related from Day 29 up to Day 387.
Groups:
- BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13); BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13); BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11); BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12); BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14): BNT162b2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection (P/B regimen), expansion cohort.
- BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B); BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B); BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B); BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B): BNT162c2: Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection P/B regimen).
Arm/Group | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/6 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/15 | 0/15 | 0/30 | 1/90 | 0/20 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/6 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 2/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 1/12 | 3/12 | 0/12 | 0/15 | 3/15 | 0/30 | 3/90 | 1/20 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 9/12 | 9/12 | 5/6 | 9/12 | 2/12 | 12/12 | 6/12 | 12/12 | 12/12 | 12/12 | 3/12 | 4/12 | 9/12 | 8/12 | 7/12 | 12/12 | 10/12 | 11/12 | 4/12 | 7/12 | 4/12 | 3/15 | 11/15 | 13/30 | 48/90 | 9/20 | 4/12 | 5/12 | 4/12 | 2/12 | 10/12 | 9/12 | 5/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg (N=12) | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg (N=12) | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg (N=6) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg (N=12) | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg (N=12) | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg (N=12) | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg (N=12) | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg (N=12) | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg (N=12) | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg (N=12) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) (N=15) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) (N=15) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) (N=30) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) (N=90) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14) (N=20) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD) (N=12)
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.1 μg (N=12) | BNT162a1 - Part A Participants Aged 18 to 55 Years - 0.3 μg (N=12) | BNT162a1 - Part A Participants Aged 18 to 55 Years - 3 μg (N=6) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 1 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 3 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 10 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 20 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 30 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 50 μg (N=12) | BNT162b1 - Part A Participants Aged 18 to 55 Years - 60 μg (N=12) | BNT162b1 - Part A Participants Aged 56 to 85 Years - 10 μg (N=12) | BNT162b1 - Part A Participants Aged 56 to 85 Years - 20 μg (N=12) | BNT162b1 - Part A Participants Aged 56 to 85 Years - 30 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 1 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 3 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 10 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 20 μg (N=12) | BNT162b2 - Part A Participants Aged 18 to 55 Years - 30 μg (N=12) | BNT162b2 - Part A Participants Aged 56 to 85 Years - 10 μg (N=12) | BNT162b2 - Part A Participants Aged 56 to 85 Years - 20 μg (N=12) | BNT162b2 - Part A Participants Aged 56 to 85 Years - 30 μg (N=12) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg HIV (Cohort 13) (N=15) | BNT162b2 - Part A IC Participants Aged 18 to 85 Years - 30 μg Post-transplant (Cohort 13) (N=15) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 3 & 30 μg (Cohort 11) (N=30) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 12) (N=90) | BNT162b2 - Part A Participants Aged 18 to 85 Years - 30 μg (Cohort 14) (N=20) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (P/B) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (P/B) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (P/B) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 3 μg (P/B) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.1 μg (SD) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.3 μg (SD) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 0.6 μg (SD) (N=12) | BNT162c2 - Part A Participants Aged 18 to 55 Years - 1 μg (SD) (N=12)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 7 | 0 | 6 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 3
Influenza like illness (General disorders) | 3 | 8 | 1 | 4 | 0 | 8 | 0 | 10 | 11 | 10 | 0 | 0 | 0 | 2 | 0 | 7 | 2 | 4 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 3 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1
Injection site reaction (General disorders) | 9 | 8 | 1 | 4 | 0 | 8 | 0 | 11 | 12 | 6 | 0 | 0 | 0 | 2 | 0 | 11 | 9 | 10 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 9
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cestode infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 5 | 0 | 8 | 1 | 8 | 5 | 2 | 1 | 0 | 1 | 0 | 1 | 4 | 2 | 1 | 1 | 2 | 3 | 0 | 2 | 3 | 10 | 2 | 1 | 1 | 1 | 0 | 4 | 3 | 1 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital discomfort (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site paraesthesia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Diastolic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site discolouration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site hypersensitivity (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site hypoaesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strength abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papilloma excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone hypertrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Physical disability (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental care (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mole excision (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT04380701/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT04380701/SAP_001.pdf